CLINICAL TRIAL: NCT01819818
Title: Korea Post-Marketing Surveillance of Invega Sustenna
Brief Title: A Study to Observe the Safety and Tolerability of Paliperidone Palmitate (Invega Sustenna) in Korean Schizophrenic Patients
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100810; R092670SCH4007 (Other: Janssen Korea, Ltd., Korea); PALM-KOR-PMS (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2013-01-18; First posted 2013-03-28 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone palmitate; Invega; Sustenna; Korea
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paliperidone palmitate
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Korean schizophrenic participants receiving paliperidone palmitate as an intramuscular injections will be observed.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of paliperidone palmitate over a 9-week period for participants with schizophrenia in Korea.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center, prospective (look forward using observations collected following participant enrollment), non-comparative, non-randomized (the study medication is not assigned by chance), study. Safety and efficacy of paliperidone palmitate will be observed in Korean schizophrenic participants for 25 weeks. Approximately 3000 participants will be observed in this study and the study duration will be 25 weeks. Safety evaluations will include assessment of adverse events, concomitant medications, physical examination, and psychiatric history.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with schizophrenia
* Participants prescribed with paliperidone palmitate for acute or maintenance treatment

Exclusion Criteria:

* Participants who received paliperidone palmitate for other than the approved indication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with schizophrenia and prescribed with paliperidone palmitate for acute or maintenance treatment.
Sampling Method: Non-Probability Sample
Enrollment: 3267 (Actual)
Dates: Start 2011-05-23 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events up to Week 9 | Up to Week 9

SECONDARY OUTCOMES:
Number of participants with adverse events up to Week 25 | Up to Week 25
Change from baseline in Clinical Global impression-Severity (CGI-S) scale scores | Baseline (Day 1), Week 5, Week 9, Week 13, Week 17, Week 21, and Week 25
  The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Change from baseline in Personal and Social Performance (PSP) scale scores | Baseline (Day 1), Week 5, Week 9, Week 13, Week 17, Week 21, and Week 25
  This PSP assesses the degree of a participants dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (i, absent to vi, very severe) in each of the 4 domains. Based on the four domains there will be one total score. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; =< 30, functioning so poorly as to require intensive supervision.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (1):
- KyungKi, South Korea